CLINICAL TRIAL: NCT07365241
Title: A Phase 3 Randomized, Open Label, Multicenter Study to Evaluate the Safety and Efficacy of ABBV-706 Versus Standard of Care in Subjects With Relapsed/Refractory Small Cell Lung Cancer (SCLC)
Brief Title: A Study to Evaluate Adverse Events and Change in Disease Activity of Intravenous ABBV-706 Versus Standard of Care in Adult Participants With Relapsed/Refractory Small Cell Lung Cancer
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M23-384; 2025-523819-11 (Other: EU CT)
Record Dates: First submitted 2026-01-22; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Small Cell Lung Cancer
Keywords: Small Cell Lung Cancer; SCLC; ABBV-706; Topotecan; Lurbinectedin; Amrubicin; Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma; Neoplasms | interventions — Topotecan; PM 01183; amrubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- ABBV-706 (Experimental): Participants will receive ABBV-706 as part of the 53 month study duration.
  Interventions: Drug: ABBV-706
- Stand of Care (SOC) (Active Comparator): Participants will receive SOC (topotecan, lurbinectedin, and amrubicin) as part of the 53 month study duration.
  Interventions: Drug: Topotecan; Drug: Lurbinectedin; Drug: Amrubicin

INTERVENTIONS:
Drug: ABBV-706 — Intravenous (IV) Infusion
  Arms: ABBV-706
Drug: Topotecan — IV Infusion
  Arms: Stand of Care (SOC)
Drug: Topotecan — Oral
  Arms: Stand of Care (SOC)
Drug: Lurbinectedin — IV Infusion
  Arms: Stand of Care (SOC)
Drug: Amrubicin — IV Infusion
  Arms: Stand of Care (SOC)

SUMMARY:
Small cell lung cancer (SCLC) is characterized by aggressive and rapid growth and a tendency to develop early spread to distant sites including mediastinal lymph nodes, liver, bones, adrenal glands, and brain. The purpose of this study is to assess safety, tolerability, and change in disease activity of ABBV-706 compared to standard of care (SOC) treatment (topotecan, lurbinectedin, or amrubicin).

ABBV-706 is an investigational drug being developed for the treatment of SCLC. There are two treatment arms in this study. Participants will either receive ABBV-706 or SOC. Approximately 531 adult participants will be enrolled in the study across 175 sites worldwide.

Participants with SCLC will receive intravenous (IV) ABBV-706 or SOC [topotecan (IV or orally), or lubinectedin (IV), or amrubicin (IV)]. The estimated duration of the study is approximately 53 months.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic and may require frequent medical assessments, blood tests, questionnaires, and scans.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of histologically or cytologically confirmed Relapsed/Refractory (R/R) Small Cell Lung Cancer (SCLC).
* Participants must have progressed on prior systemic therapy, with CPI (if eligible) and prior tarlatamab, defined as:

  * In the 1L and 2L setting respectively, platinum-based chemotherapy (i.e., carboplatin or cisplatin and etoposide with CPI, if eligible for CPI) and 2L tarlatamab; or
  * In the 1L and 2L setting, platinum-based chemotherapy (i.e., carboplatin and etoposide with atezolizumab and lurbinectedin in combination with atezolizumab maintenance and 2L tarlatamab; or
  * In the 1L setting, platinum-based chemotherapy (i.e., carboplatin or cisplatin and etoposide with CPI if eligible) in combination with tarlatamab in frontline induction and/or maintenance
* Participants must be considered suitable to receive SOC comparator (topotecan, lurbinectedin, or amrubicin).
* Participants must have an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 1 during the screening period prior to the first dose of study treatment.
* Participants must have measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. Target lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
* Participants with brain metastasis from an extracranial solid tumor are eligible if the brain metastases are:

  * Previously treated and not requiring anticonvulsants and steroids for at least 7 days prior to first dose of study treatment. If required for management, subjects on a steroid equivalent of prednisone dose of ≤ 10 mg/day are eligible or;
  * Untreated and asymptomatic not requiring anticonvulsants and steroids for at least 7 days prior to the first dose of study treatment. If required for management, subjects on a steroid equivalent of prednisone of ≤ 10 mg/day are eligible.

Exclusion Criteria:

* Participants with known active/symptomatic central nervous system metastases.
* Participants with a history of interstitial lung disease (ILD) or pneumonitis that previously required treatment with systemic steroids, or any evidence of active ILD/pneumonitis on screening chest computed tomography (CT) scan.
* Participants with any clinically significant conditions that would adversely affect the participation in the study, and the subject should have a life expectancy of at least 3 months.
* Participants who have received prior treatment with a seizure-related 6 homolog (SEZ6) targeted Antibody drug conjugate (ADC), other targeted ADCs, or any other investigational agent not including tarlatamab in 1L.
* Participants who have received prior treatment with any Top1i such as topotecan, irinotecan, belotecan, camptothecin, rubitecan, exatecan or locally approved topoisomerase I inhibitor (Top1i) payload.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 531 (Estimated)
Dates: Start 2026-04-14 (Estimated); Primary Completion 2030-09 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Objective Response (OR) as Measured by Overall Response Rate (ORR) Based on Blinded Independent Central Review (BICR) | Up to approximately 24 months
  OR is defined as participants achieving a best overall response (BOR) of confirmed complete response (CR)/partial response (PR) per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 as determined by BICR assessment prior to initiation of subsequent anti-cancer therapy. OR will be summarized by ORR, defined as the percentage of participants achieving OR and will be summarized for each arm with its associated 95% confidence interval (CI).
Overall Survival (OS) | Up to approximately 28 months
  OS is defined as the time from the date of randomization to the date of death of any cause.

SECONDARY OUTCOMES:
Progression-free survival (PFS) based on BICR assessment per RECIST v1.1. | Up to Approximately 24 Months
  PFS is defined as the time from the date of randomization to the first documentation of radiographic disease progression per RECIST v1.1 based on BICR assessment or death from any cause, whichever occurs first.
Duration of response (DoR) based on BICR assessment per RECIST v1.1. | Up to Approximately 24 Months
  DoR is defined as the time from the initial response of confirmed CR or PR per RECIST v1.1 based on BICR assessment to radiographic disease progression per RECIST v1.1 based on BICR assessment, or death of any cause, whichever occurs first.
Change from baseline at Week 12 in physical functioning as measured by the physical functioning domain of the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30). | Week 12
  Health-related quality-of-life (HRQoL) and symptoms will be assessed with the EORTC QLQ-C30, version 3.0. The EORTC QLQ-C30 is a 30-item patient-reported questionnaire composed of both multi-item and single scales including 5 functional scales (physical, role, emotional, social, and cognitive), 3 symptom scales (fatigue, nausea and vomiting, and pain), a global health status (GHS)/QoL scale, and 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). Participants rate items on a 4 point scale ranging from 1 to 4 (1 = Not at All, 2 = A Little, 3 = Quite a Bit, and 4 = Very Much).
Change from baseline at Week 12 in Global Health Status (GHS)/Quality of life (QoL) as measured by the EORTC QLQ-C30 GHS/QoL scale | Week 12
  Health-related quality-of-life and symptoms will be assessed with the EORTC QLQ-C30, version 3.0. The EORTC QLQ-C30 is a 30-item patient-reported questionnaire composed of both multi-item and single scales including 5 functional scales (physical, role, emotional, social, and cognitive), 3 symptom scales (fatigue, nausea and vomiting, and pain), a GHS/QoL scale, and 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). Participants rate items on a 4 point scale ranging from 1 to 4 (1 = Not at All, 2 = A Little, 3 = Quite a Bit, and 4 = Very Much).
Number of Participants with Adverse Events (AEs) | Up to Approximately 53 Months
  An AE is defined as any untoward medical occurrence in a patient or clinical investigation in which a participant is administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing, visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M23-384